CLINICAL TRIAL: NCT02777229
Title: A Phase III Randomized, Open Label Trial to Evaluate Dolutegravir Versus Efavirenz 400 mg, Both Combined With Tenofovir Disoproxil Fumarate + Lamivudine for the Initial Management of HIV Infected Adults in Resource-limited Settings
Brief Title: Efficacy and Safety of a Dolutegravir-based Regimen for the Initial Management of HIV Infected Adults in Resource-limited Settings
Acronym: NAMSAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: Institut de Recherche pour le Developpement (Other Government); UNITAID (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS 12313 NAMSAL
Record Dates: First submitted 2016-03-01; First posted 2016-05-19 (Estimated); Last update posted 2021-08-31 (Actual); Status verified 2021-02

CONDITIONS: HIV-1 Infection
Keywords: Dolutegravir; Efavirenz-low-dose
MeSH Terms: interventions — dolutegravir; Tenofovir; Lamivudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dolutegravir (Experimental): Dolutegravir 50 mg Quaque die (QD) + tenofovir disoproxil fumarate/lamivudine 300 mg/ 300 mg Fixed Dose Combination (FDC) QD
  Interventions: Drug: Dolutegravir 50 mg; Drug: Tenofovir disoproxil fumarate 300 mg / lamivudine 300 mg
- Efavirenz (Active Comparator): Efavirenz 400 mg QD + tenofovir disoproxil fumarate/lamivudine 300 mg/ 300 mg FDC QD
  Interventions: Drug: Tenofovir disoproxil fumarate 300 mg / lamivudine 300 mg; Drug: Efavirenz 400 mg

INTERVENTIONS:
Drug: Dolutegravir 50 mg — 1 tablet once a day
  Other Names: DTG
  Arms: Dolutegravir
Drug: Tenofovir disoproxil fumarate 300 mg / lamivudine 300 mg — Fixed dose combination, 1 tablet once a day
  Other Names: TDF / 3TC
Drug: Efavirenz 400 mg — 1 tablets once a day
  Other Names: EFV400
  Arms: Efavirenz

SUMMARY:
Several reports indicate that treatment failure due to HIV resistance or to adverse event-related discontinuation could compromise the effectiveness of scaling-up antiretroviral treatment (ART), especially when lack of access to viral load is a concern. Combined with other nucleoside reverse transcriptase inhibitor, Dolutegravir (DTG) is a very promising alternative to the current first-line non nucleoside reverse transcriptase inhibitor-based regimens.

Initial evaluations of DTG conducted in high income countries showed excellent efficacy and safety and indicated high genetic barrier thus preserving second line treatment. As a consequence, DTG-based regimens have been recently included in the first-line options in the national guidelines for ART of several high-income countries. However, the clinical trials evaluating DTG-based regimens have been conducted in highly controlled conditions, including baseline resistance testing and regular viral load monitoring. Moreover, these trials included a high proportion of men with rare co-morbidities.

There is need to evaluate how a DTG-based regimen will perform in real-world conditions within resources-constrained settings, where viral load monitoring is limited, and where the majority of HIV patients are women with important family planning consideration and NAMSAL trial is a randomized clinical trial which aims to evaluate efficacy and safety over 48, 96 and 192 weeks of DTG + tenofovir disoproxil fumarate/lamivudine versus Efavirenz (EFV) + tenofovir disoproxil fumarate/lamivudine in 606 ART-naïve HIV-1-infected adults in Cameroon. A set of efficacy and safety endpoints will be compared over 48, 96 and 192 weeks between the two arms including the proportion of patients with viral load <50 copies/mL and incidence of severe adverse events.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Age ≥ 18 years
* Abtiretroviral-naïve, including above 7 days of cumulative prior antiretroviral therapy at any time prior to study entry.
* For women of childbearing potential: acceptance to use effective contraceptive methods
* Provision of written informed consent

Exclusion Criteria:

* Infection with HIV-1 group O, N, P
* Infection or co-infection with HIV-2
* Absolute neutrophil count (ANC) < 500 cells/mm3
* Hemoglobin < 7.0 g/dL
* Platelet count < 50,000 cells/mm3
* AST and/or ALT > 5 x Upper Limit of Normal (ULN)
* Calculated creatinine clearance < 50 mL/min
* Active opportunistic or severe disease not under adequate control
* For women of childbearing age : Pregnancy/breastfeeding
* History or presence of allergy and/or contraindications to the trial drugs or their components
* Severe psychiatric illness
* Severe hepatic failure Patients co-infected with tuberculosis (TB), receiving a TB treatment and with stable clinical condition will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with Viral Load (VL) <50 cp/mL | week 48
  Proportion of patients with Viral Load (VL) <50 cp/mL at week 48 (FDA snapshot algorithm)

SECONDARY OUTCOMES:
Proportion of patients with Viral Load (VL) <50 cp/mL | week 96
  Proportion of patients with Viral Load (VL) <50 cp/mL at week 96 (FDA snapshot algorithm)
Proportion of patients with Viral Load (VL) <50 cp/mL | week 24
  Proportion of patients with VL< 50 cp/mL at week 24 (FDA snapshot algorithm)
Proportion of patients with Viral Load (VL) < 200 cp/mL | week 24, week 48, week 96, week 144, week 192
  Proportion of patients with VL< 200 cp/mL (FDA snapshot algorithm)
Time to virologic failure | week 48, week 96, week 144, week 192
  Time to virologic failure
Changes in Cluster of differentiation 4 (CD4)-cell count from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in Cluster of differentiation 4 (CD4)-cell count from baseline to endpoints week-48, -96, -144, -192
Time to death or to disease progression | week 48, week 96, week 144, week 192
  Time to death or to disease progression
Time to first toxicity failure | week 48, week 96, week 144, week 192
  Time to first toxicity failure
Incidence of first grade 3 or 4 clinical adverse event | week 48, week 96, week 144, week 192
  Incidence of first grade 3 or 4 clinical adverse event
Incidence of first grade 3 or 4 laboratory adverse event | week 48, week 96, week 144, week 192
  Incidence of first grade 3 or 4 laboratory adverse event
AE and SAE | week 48, week 96, week 144, week 192
  Incidence of adverse events (AE) and serious adverse event (SAE)
Time to treatment discontinuation | week 48, week 96, week 144, week 192
  Time to treatment discontinuation
Hemoglobine changes from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in hemoglobin Time to virologic failure from baseline to endpoints week-48, -96, -144, -192
Changes in creatinine from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in creatinine from baseline to endpoints week-48, -96, -144, -192
Changes in estimated glomerular filtration rate from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in estimated glomerular filtration rate from baseline to endpoints week-48, -96, -144, -192
Changes in Aspartate Aminotransferase (AST) ffrom baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in Aspartate Aminotransferase (AST) from baseline to endpoints week-48, -96, -144, -192
Changes in Alanine Aminotransferase (ALT) from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in Alanine Aminotransferase (ALT) from baseline to endpoints week-48, -96, -144, -192
Changes in level of fasting glucose from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in level of fasting glucose from baseline to endpoints week-48, -96, -144, -192
Changes in level of total cholesterol from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in level of total cholesterol from baseline to endpoints week-48, -96, -144, -192
Changes in level of triglycerides from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in level of triglycerides from baseline to endpoints week-48, -96, -144, -192
Changes in level of HDL from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Changes in level of HDL from baseline to endpoints week-48, -96, -144, -192
Proportion of patients defaulting clinic schedule | week 48, week 96, week 144, week 192
  Proportion of patients defaulting clinic schedule
Mean medication adherence level from baseline to endpoints week-48, -96, -144, -192 | week 48, week 96, week 144, week 192
  Mean medication adherence level from baseline to endpoints week-48, -96, -144, -192
Mean change in Depression Anxiety Stress Scale from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Mean change in Depression Anxiety Stress Scale from baseline to endpoints week-48, -96, -144, -192
  * Depression Normal 0-9, Mild 10-13, Moderate 14-20, Severe 21-27, Extremely Severe +28
  * Anxiety Normal 0-7, Mild 8-9, Moderate 10-14, Severe 15-19, Extremely Severe +20
  * Stress Normal 0-14, Mild 15-18, Moderate 19-25, Severe 26-33, Extremely Severe +34
Mean change in Quality of life score assessed by the Short Form health survey from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96, week 144, week 192
  Mean change in Quality of life score assessed by the Short Form health survey from baseline to endpoints week-48, -96, -144, -192 (Score varies according to the items, in order to test the vigilance of the patient. Reading the results provides a semantic appreciation)
Mean change in EFV-related symptoms questionnaire score from baseline to endpoints week-48, -96, -144, -192 | Baseline, week 48, week 96
  Mean change in EFV-related symptoms questionnaire score from baseline to endpoints week-48, -96, -144, -192
Tobacco status consumtion | week 192
  The status of tobacco smoker / non-smoker will be requested.
HbA1c | week 192
  Levels of glycated hemoglobin
hsPCR | week 192
  Levels of high sensitivity protein C reactive
Lipodistrophia | week 192
  Qualitative and quantitative measurements of soft tissue composition = Lipodistrophia
CIMT | week 192
  Mesures of Carotid Intima-Media Thickness
PWV | week 192
  Mesures of Pulse Wave Velocity
Levels of adiponectin | Baseline, week 48, week 96, week 144, week 192
  Levels of adiponectin
Levels of leptin | Baseline, week 48, week 96, week 144, week 192
  Levels of leptin
Levels of ghrelin | Baseline, week 48, week 96, week 144, week 192
  Levels of ghrelin

CONTACTS AND LOCATIONS:
Overall Officials: Eric Delaporte, MD, PhD, Principal Investigator — IRD, INSERM, University Montpellier; Charles Kouanfack, MD, PhD, Principal Investigator — Central Hospital
Locations (3):
- Cameroon (3):
  - Cité verte Hospital, Yaoundé
  - Hopital Central, Yaoundé
  - Military Hospital, Yaoundé

REFERENCES:
- [Derived] Mpoudi-Etame M, Tovar Sanchez T, Bousmah MA, Omgba Bassega P, Olinga J, Mimbe E, Foalem M, Chiep C, Edimo S, Varloteaux M, Pelloquin R, Lamare N, Boyer S, Peeters M, Reynes J, Calmy A, Hill A, Delaporte E, Kouanfack C; New Antiretroviral and Monitoring Strategies in HIV-infected Adults in Low-income countries (NAMSAL-ANRS-12313) study group. Durability of the Efficacy and Safety of Dolutegravir-Based and Low-Dose Efavirenz-Based Regimens for the Initial Treatment of Human Immunodeficiency Virus Type 1 Infection in Cameroon: Week 192 Data of the NAMSAL-ANRS-12313 Study. Open Forum Infect Dis. 2023 Nov 20;10(12):ofad582. doi: 10.1093/ofid/ofad582. eCollection 2023 Dec. PMID 38156046
- [Derived] Bousmah MA, Protopopescu C, Mpoudi-Etame M, Omgba Bassega P, Maradan G, Olinga J, Varloteaux M, Tovar-Sanchez T, Delaporte E, Kouanfack C, Boyer S; NAMSAL ANRS 12313 Study Group. Improvements in Patient-Reported Outcomes Following Initiation of Dolutegravir-Based or Low-Dose Efavirenz-Based First-Line Antiretroviral Therapy: A Four-Year Longitudinal Analysis in Cameroon (NAMSAL ANRS 12313 Trial). J Acquir Immune Defic Syndr. 2023 Nov 1;94(3):262-272. doi: 10.1097/QAI.0000000000003273. PMID 37851566
- [Derived] Bousmah MA, Nishimwe ML, Tovar-Sanchez T, Lantche Wandji M, Mpoudi-Etame M, Maradan G, Omgba Bassega P, Varloteaux M, Montoyo A, Kouanfack C, Delaporte E, Boyer S; New Antiretroviral and Monitoring Strategies in HIV-infected Adults in Low-Income Countries (NAMSAL) ANRS 12313 Study Group. Cost-Utility Analysis of a Dolutegravir-Based Versus Low-Dose Efavirenz-Based Regimen for the Initial Treatment of HIV-Infected Patients in Cameroon (NAMSAL ANRS 12313 Trial). Pharmacoeconomics. 2021 Mar;39(3):331-343. doi: 10.1007/s40273-020-00987-3. Epub 2020 Dec 23. PMID 33355914
- [Derived] Calmy A, Tovar Sanchez T, Kouanfack C, Mpoudi-Etame M, Leroy S, Perrineau S, Lantche Wandji M, Tetsa Tata D, Omgba Bassega P, Abong Bwenda T, Varloteaux M, Tongo M, Mpoudi-Ngole E, Montoyo A, Mercier N, LeMoing V, Peeters M, Reynes J, Delaporte E; New Antiretroviral and Monitoring Strategies in HIV-infected Adults in Low-Income Countries (NAMSAL) ANRS 12313 Study Group. Dolutegravir-based and low-dose efavirenz-based regimen for the initial treatment of HIV-1 infection (NAMSAL): week 96 results from a two-group, multicentre, randomised, open label, phase 3 non-inferiority trial in Cameroon. Lancet HIV. 2020 Oct;7(10):e677-e687. doi: 10.1016/S2352-3018(20)30238-1. PMID 33010241
- [Derived] NAMSAL ANRS 12313 Study Group; Kouanfack C, Mpoudi-Etame M, Omgba Bassega P, Eymard-Duvernay S, Leroy S, Boyer S, Peeters M, Calmy A, Delaporte E. Dolutegravir-Based or Low-Dose Efavirenz-Based Regimen for the Treatment of HIV-1. N Engl J Med. 2019 Aug 29;381(9):816-826. doi: 10.1056/NEJMoa1904340. Epub 2019 Jul 24. PMID 31339676